CLINICAL TRIAL: NCT06193967
Title: Enhancing Child Digital Dietary Self-monitoring: Proof-of-concept Trial
Brief Title: Enhancing Child Dietary Self-monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Executive Associate Dean of Research & Operations, College of Education, Health, and Human Sciences, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: UTK IRB-23-07903-XP
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BASIC (No Intervention): Children will be asked to track their intake of fruits, vegetables, sweet and salty snack foods, and sugary drinks in the web-based dietary self-monitoring (DSM) log for 4 weeks. Each child will be provided with a personal URL to access their log, which can be accessed from any internet-capable device (computer, phone, etc.). Caregivers will be asked to review their child's log each day and complete a caregiver check-in in the DSM log.
- PRAISE (Experimental): In addition to conditions of the BASIC group, caregivers will also be asked to provide praise to their child for engaging in DSM over the 4 weeks. Additionally, when the caregiver completes caregiver check-ins in the DSM log, they will receive a prompt to also complete a praise check-in.
  Interventions: Behavioral: Caregiver Praise
- GAME (Experimental): In addition to the conditions of the BASIC group, the child's log will also include a virtual pet that evolves over time as he/she uses the log. As the child earns points, the pet will level up and grow over time.
  Interventions: Behavioral: Gamification
- PRAISE+GAME (Experimental): In addition to conditions of the BASIC group, caregivers will also be asked to provide praise to their child for engaging in DSM over the 4 weeks. Additionally, when the caregiver completes caregiver check-ins in the DSM log, they will receive a prompt to also complete a praise check-in. The child's log will also include a virtual pet that evolves over time as he/she uses the log. As the child earns points, the pet will level up and grow over time.
  Interventions: Behavioral: Caregiver Praise; Behavioral: Gamification

INTERVENTIONS:
Behavioral: Caregiver Praise — Caregivers will provide praise for child's engagement in dietary self-monitoring behaviors as a form of positive reinforcement
  Arms: PRAISE; PRAISE+GAME
Behavioral: Gamification — DSM logs will include gamification (points, levels, virtual pets) as positive reinforcement for child's engagement in dietary self-monitoring behaviors
  Arms: GAME; PRAISE+GAME

SUMMARY:
The goal of this clinical trial was to test the preliminary efficacy of a digital dietary self-monitoring (dDSM) log that uses positive reinforcement strategies (caregiver praise and gamification) to improve child engagement in DSM. The main aims were to:

* Conduct a proof-of-concept trial that examines the effects of positive reinforcement on child DSM behaviors.
* Explore differences in children's intrinsic motivation.

Participating children will be instructed to self-monitor their daily intake of targeted food groups (fruits, vegetables, sweet and salty snack foods, and sugar-sweetened beverages) for 4 weeks using a personal web-based DSM log. Each child-caregiver dyad will be randomly assigned to 1 of 4 conditions: BASIC, PRAISE, GAME, or PRAISE+GAME. For PRAISE and PRAISE+GAME conditions, caregivers will be instructed to provide daily process praise to their child related to DSM behaviors. For GAME and PRAISE+GAME conditions, logs will integrate three game mechanics: points, levels, and a virtual pet. Points will be accumulated for engaging in DSM behaviors, and accrual of points will evolve a virtual pet over time.

DETAILED DESCRIPTION:
The objective of the proposed study was to test the usability, acceptability, and preliminary efficacy of a digital dietary self-monitoring (dDSM) log that used positive reinforcement strategies (caregiver praise and gamification) to improve child engagement in DSM.

For this proof of concept trial, a mobile-optimized, web-based dDSM log was developed to test the two positive reinforcement strategies: caregiver praise and gamification. The dDSM log was developed as a mobile-optimized website, rather than an app, so that phone operating systems were not a limitation of use. Families were therefore able to access the dDSM log from a computer, smartphone, or other internet-enabled device. All dDSM logs included three basic features: 1) the ability to log targeted food groups with amounts and servings consumed, 2) the ability to indicate logging was complete for the day, and 3) access to a help feature that provided guidance on tracking and serving sizes. Children were instructed to self-monitor their daily intake of the following food groups: fruits, vegetables, sweet and salty snack foods, and sugar-sweetened beverages (SSBs). DSM focused on these four food groups because they had an established influence on health. Fruit and vegetable consumption was associated with a decreased risk of chronic disease, and reduced consumption of energy-dense foods like sweet and salty snacks and SSBs was recommended for weight loss in children. Additionally, these food groups were frequently targeted in childhood obesity treatment and were easily understood by young children.

Using a 2x2 factorial design, each child-caregiver dyad was randomly assigned to 1 of 4 conditions: BASIC, PRAISE, GAME, or PRAISE+GAME. Each child was provided a unique URL to access a personal dDSM log with the appropriate, randomly assigned features (praise and/or gamification). For PRAISE and PRAISE+GAME conditions, caregivers were instructed to provide daily process praise to their child related to DSM behaviors. While DSM was frequently implemented within treatment, children in the proposed study engaged in DSM without a concurrent intervention to tightly control the influence of the independent variables on DSM behaviors only (as compared to having all adult caregivers learn how to praise or having caregivers focus their praise on achieving dietary goals, which were both standard components of family-based childhood obesity interventions). Thus, only caregivers randomized to PRAISE or PRAISE+GAME were instructed on praise and, in the absence of dietary goals for intervention, caregivers had only one behavior (DSM) to praise. For GAME and PRAISE+GAME conditions, logs integrated three game mechanics: points, levels, and a virtual pet. Points were accumulated for engaging in DSM behaviors, and the accrual of points evolved a virtual pet over time, acting as a digital token economy. The number of points to level up increased with each level, so that each consecutive level was harder to attain than the previous one. At the end of the 4-week DSM period, families who completed follow-up assessments received two $25 gift cards (one for the caregiver, one for the child) and were provided access to a short online behavioral nutrition education program.

The primary DSM outcomes were frequency (i.e., the number of days any food/beverage item was tracked or logging was marked complete) and timing (i.e., how many sessions of recording were completed each day and whether foods/beverages were logged on the day of intake). On days in which no targeted food group was consumed, children had the ability to mark logging as complete for the day (Figure 1a). Indicating logging was complete in the absence of any tracked foods was considered a "tracked" day. Pre-post changes in intrinsic motivation were also examined.

ELIGIBILITY:
Inclusion Criteria:

* Families with children ages 8-12 years with body mass index (BMI)-for-age ≥ 5th percentile who report eating foods/beverages (any serving size) from ≥2 targeted food groups (fruits, vegetables, sweet and salty snack foods, and SSBs) on ≥3 days/week each and who have an adult caregiver ≥18 years of age willing to participate
* Family has reliable access to the internet via phone, computer, or another device that the child is able and permitted to operate

Exclusion Criteria:

* Child has major psychiatric diseases or organic brain syndromes
* Family does not live in the greater Knoxville area
* Family does not speak English

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Germann JN, Kirschenbaum DS, Rich BH. Child and parental self-monitoring as determinants of success in the treatment of morbid obesity in low-income minority children. J Pediatr Psychol. 2007 Jan-Feb;32(1):111-21. doi: 10.1093/jpepsy/jsl007. Epub 2006 Jun 14. PMID 16775083
- [Background] Mockus DS, Macera CA, Wingard DL, Peddecord M, Thomas RG, Wilfley DE. Dietary self-monitoring and its impact on weight loss in overweight children. Int J Pediatr Obes. 2011 Aug;6(3-4):197-205. doi: 10.3109/17477166.2011.590196. Epub 2011 Jul 4. PMID 21722068
- [Background] Saelens BE, McGrath AM. Self-monitoring adherence and adolescent weight control efficacy. Children's Health Care. 2003;32(2):137-152.
- [Background] Dalle Grave R, Centis E, Marzocchi R, El Ghoch M, Marchesini G. Major factors for facilitating change in behavioral strategies to reduce obesity. Psychol Res Behav Manag. 2013 Oct 3;6:101-10. doi: 10.2147/PRBM.S40460. PMID 24124398
- [Background] Guideline Development Panel for Treatment of Obesity, American Psychological Association. Summary of the clinical practice guideline for multicomponent behavioral treatment of obesity and overweight in children and adolescents. Am Psychol. 2020 Feb-Mar;75(2):178-188. doi: 10.1037/amp0000530. PMID 32052993
- [Background] Favell JE. The power of positive reinforcement: a handbook of behavior modification. Charles C Thomas; 1977.
- [Background] Griffiths LA, Douglas SM, Raynor HA. The role of structure in dietary approaches for the treatment of pediatric overweight and obesity: A critical review. Obes Rev. 2021 Sep;22(9):e13266. doi: 10.1111/obr.13266. Epub 2021 May 5. PMID 33955110
- [Background] Henggeler SW, Sheidow AJ. Empirically supported family-based treatments for conduct disorder and delinquency in adolescents. J Marital Fam Ther. 2012 Jan;38(1):30-58. doi: 10.1111/j.1752-0606.2011.00244.x. Epub 2011 Sep 20. PMID 22283380
- [Background] Freeman JB, Garcia AM. Family based treatment for young children with OCD: therapist guide. Oxford University Press; 2008.
- [Background] Garett R, Young SD. Health care gamification: a study of game mechanics and elements. Technology, Knowledge and Learning. 2019;24(3):341-353.
- [Background] Kumar VS, Wentzell KJ, Mikkelsen T, Pentland A, Laffel LM. The DAILY (Daily Automated Intensive Log for Youth) trial: a wireless, portable system to improve adherence and glycemic control in youth with diabetes. Diabetes Technol Ther. 2004 Aug;6(4):445-53. doi: 10.1089/1520915041705893. PMID 15320998
- [Background] Cafazzo JA, Casselman M, Hamming N, Katzman DK, Palmert MR. Design of an mHealth app for the self-management of adolescent type 1 diabetes: a pilot study. J Med Internet Res. 2012 May 8;14(3):e70. doi: 10.2196/jmir.2058. PMID 22564332
- [Background] Klingensmith GJ, Aisenberg J, Kaufman F, Halvorson M, Cruz E, Riordan ME, Varma C, Pardo S, Viggiani MT, Wallace JF, Schachner HC, Bailey T. Evaluation of a combined blood glucose monitoring and gaming system (Didget(R)) for motivation in children, adolescents, and young adults with type 1 diabetes. Pediatr Diabetes. 2013 Aug;14(5):350-7. doi: 10.1111/j.1399-5448.2011.00791.x. Epub 2011 Jun 23. PMID 21699639
- [Background] Swartwout E, El-Zein A, Deyo P, Sweenie R, Streisand R. Use of Gaming in Self-Management of Diabetes in Teens. Curr Diab Rep. 2016 Jul;16(7):59. doi: 10.1007/s11892-016-0754-2. PMID 27155609
- [Background] Debong F, Mayer H, Kober J. Real-World Assessments of mySugr Mobile Health App. Diabetes Technol Ther. 2019 Jun;21(S2):S235-S240. doi: 10.1089/dia.2019.0019. PMID 31169427
- [Background] Deci EL, Koestner R, Ryan RM. A meta-analytic review of experiments examining the effects of extrinsic rewards on intrinsic motivation. Psychol Bull. 1999 Nov;125(6):627-68; discussion 692-700. doi: 10.1037/0033-2909.125.6.627. PMID 10589297
- [Background] Mekler ED, Brühlmann F, Opwis K, Tuch AN. Do points, levels and leaderboards harm intrinsic motivation? An empirical analysis of common gamification elements. 2013:66-73.
- [Background] Linehan C, Kirman B, Roche B. Gamification as behavioral psychology. The Gameful world: Approaches, Issues, Applications. MIT Press; 2015:81-105.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Numbers for Protocol Enrollment, Number Started, and Number Completed reflect dyads
Period: Overall Study
Arm/Group | BASIC | PRAISE | GAME | PRAISE+GAME
Started (Dyads) | 5 | 5 | 5 | 4
Children | 5 | 5 | 5 | 4
Caregivers | 5 | 5 | 5 | 4
Completed (Dyads) | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Numbers include both child and caregiver participants
Groups:
- Total: Total of all reporting groups
Arm/Group | BASIC | PRAISE | GAME | PRAISE+GAME | Total
Number analyzed (Participants) | 10 | 10 | 10 | 8 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] — Child age Population: Child only measure
  years
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    (all) | 7.7 (4.0) | 9.2 (1.1) | 10.8 (1.3) | 9.3 (1.3) | 9.1 (2.6)
Age, Continuous [Mean (Standard Deviation); unit: years] — Caregiver age Population: Caregiver only measure
  years
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    (all) | 43.0 (2.6) | 43.0 (7.1) | 44.0 (3.6) | 41.0 (6.7) | 42.8 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Child sex Population: Child only measure
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    Female | 4 | 2 | 3 | 2 | 11
    Male | 1 | 3 | 2 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants] — Caregiver sex Population: Caregiver only measure
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    Female | 3 | 3 | 5 | 4 | 15
    Male | 2 | 2 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Child ethnicity Population: Child only measure
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    Hispanic or Latino | 1 | 0 | 0 | 0 | 1
    Not Hispanic or Latino | 4 | 5 | 5 | 4 | 18
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Caregiver ethnicity Population: Caregiver only measure
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 5 | 5 | 5 | 4 | 19
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Child race Population: Child only measure
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 1 | 1
    White | 4 | 3 | 5 | 2 | 14
    More than one race | 1 | 1 | 0 | 1 | 3
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Caregiver race Population: Caregiver only measure
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 1 | 1
    White | 5 | 3 | 5 | 2 | 15
    More than one race | 0 | 1 | 0 | 1 | 2
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Child BMI Percentile [Mean (Standard Deviation); unit: percentile] — Population: Child only measure
  percentile
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    (all) | 37.0 (17.8) | 76.8 (30.9) | 68.6 (33.7) | 60.0 (31.8) | 60.6 (30.8)
Caregiver marital status [Count of Participants; unit: Participants] — Population: Caregiver only measure
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    Married | 5 | 5 | 4 | 3 | 17
    Never married | 0 | 0 | 1 | 0 | 1
    Refused to answer | 0 | 0 | 0 | 1 | 1
Caregiver education level [Count of Participants; unit: Participants] — Population: Caregiver only measure
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    Grade 12 or GED (high school graduate) | 0 | 1 | 0 | 0 | 1
    College 1 year to 3 years (some college or technical school) | 0 | 0 | 1 | 0 | 1
    College 4 years or more (college graduate) | 5 | 4 | 4 | 4 | 17
Household income [Count of Participants; unit: Participants] — Population: Caregiver only measure
  Participants
    number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    Less than $10,000 | 0 | 0 | 0 | 0 | 0
    $10,000 to $19,999 | 0 | 0 | 0 | 0 | 0
    $20,000 to $29,999 | 0 | 0 | 1 | 0 | 1
    $30,000 to $39,999 | 0 | 0 | 0 | 0 | 0
    $40,000 to $49,999 | 0 | 0 | 0 | 0 | 0
    $50,000 to $59,999 | 0 | 0 | 0 | 0 | 0
    $60,000 to $69,999 | 0 | 1 | 0 | 0 | 1
    $70,000 to $79,999 | 0 | 0 | 0 | 1 | 1
    $80,000 to $89,999 | 0 | 0 | 0 | 0 | 0
    $90,000 to $99,999 | 0 | 0 | 0 | 0 | 0
    $100,000 to $149,999 | 0 | 1 | 1 | 2 | 4
    $150,000 or more | 5 | 3 | 3 | 1 | 12
Caregiver Parenting Styles & Dimensions Questionnaire (PSDQ) score [Mean (Standard Deviation); unit: units on a scale] — The scale for each domain is 1 to 5. A lower score indicates less adherence to the respective parenting style, while a higher score indicates greater adherence to the respective parenting style. Population: Caregiver only measure
  units on a scale
    Authoritative domain: number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    Authoritative domain | 4.1 (0.1) | 4.2 (0.5) | 4.1 (0.2) | 4.2 (0.3) | 4.1 (0.3)
    Authoritarian domain: number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    Authoritarian domain | 1.5 (0.2) | 1.5 (0.3) | 1.8 (0.3) | 1.7 (0.5) | 1.6 (0.3)
    Permissive domain: number analyzed (Participants) | 5 | 5 | 5 | 4 | 19
    Permissive domain | 2.0 (0.6) | 2.1 (0.7) | 2.6 (0.7) | 2.0 (0.3) | 2.2 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Dietary Self-monitoring Frequency, Overall
Description: I.e., number of days with any logging. DSM frequency has been shown to predict success in family-based based childhood overweight and obesity programs. A day will be counted as "tracked" if any food or beverage is logged on that day or, if no food or beverage is logged, the "Logging Complete" button is clicked.
Time Frame: 4 weeks
Population: Dyads were randomized by condition (BASIC, PRAISE, GAME, or PRAISE+GAME). However, factorial analysis was used to calculate the main effects of the independent variables, i.e. assignment to praise and assignment to gamification. Therefore, the table presents results for the same 19 enrolled children twice: 1) as assigned to praise versus not assigned to praise and 2) as assigned to gamification versus not assigned to gamification.
Measure: Mean (Standard Error); unit: days
Groups:
- No Caregiver Praise: Children not assigned to receive caregiver praise (i.e., participants from BASIC and GAME)
- Caregiver Praise: Children assigned to receive caregiver praise (i.e., participants from PRAISE and PRAISE+GAME)
- No Gamification: Children not assigned to receive gamification (i.e., participants from BASIC and PRAISE)
- Gamification: Children assigned to receive gamification (i.e., participants from GAME and PRAISE+GAME)
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
days | 23.0 (1.4) | 24.3 (1.4) | 22.0 (1.3) | 25.3 (1.4)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise; A standard alpha level of ≥ 0.05 was used to determine statistical significance; Test type: Other; p > 0.05, ANOVA; To determine the main effects of positive reinforcement on DSM behavior, a 2x2 factorial ANOVA was conducted with gamification and caregiver praise status as the independent variables and a dependent variable of DSM frequency (number of days with tracking). A gamification*caregiver praise interaction term was also included in the model to test for interactive effects
Statistical Analysis 2: Comparison: No Gamification vs Gamification; Test type: Other; p > 0.05, ANOVA; [other analysis details as in outcome 1, analysis 1]

2. Primary Outcome: Dietary Self-monitoring Frequency, Weekly
Description: I.e., number of days with any logging per week
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
days
  Week 1 | 6.8 (0.1) | 6.8 (0.1) | 6.7 (0.1) | 6.9 (0.1)
  Week 2 | 6.0 (0.4) | 6.5 (0.4) | 5.9 (0.4) | 6.6 (0.4)
  Week 3 | 5.4 (0.5) | 6.5 (0.5) | 5.4 (0.5) | 6.5 (0.5)
  Week 4 | 4.8 (0.7) | 4.6 (0.8) | 4.0 (0.7) | 5.4 (0.8)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise vs No Gamification vs Gamification; A standard alpha level of ≥ 0.05 was used to determine statistical significance; Test type: Other; p < 0.001, ANOVA; Linear mixed-factor ANOVA was used with between-subject factors of praise and gamification status, a within-subject factor of time (week), and a dependent variable of DSM frequency. Results reflect outcomes for main effect of time

3. Primary Outcome: Proportion of Items Tracked on Day of Intake, Overall
Description: Proportion of food/beverage items that were tracked on the day of intake across the 4-week DSM period
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: proportion of items tracked
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
proportion of items tracked | 0.73 (0.05) | 0.69 (0.06) | 0.70 (0.05) | 0.73 (0.06)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise; A standard alpha level of ≥ 0.05 was used to determine statistical significance; Test type: Superiority; p > 0.05, ANOVA; To determine the main effects of positive reinforcement on DSM behavior, a 2x2 factorial ANOVA was conducted with gamification and caregiver praise status as the independent variables and a dependent variable of DSM timing (proportion of items tracked on day of intake). A gamification*caregiver praise interaction term was also included in the model to test for interactive effects
Statistical Analysis 2: Comparison: No Gamification vs Gamification; Test type: Other; p > 0.05, ANOVA; [other analysis details as in outcome 3, analysis 1]

4. Primary Outcome: Proportion of Items Tracked on Day of Intake, Weekly
Description: Proportion of food/beverage items that were tracked on the day of intake by week
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: proportion of items tracked
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
proportion of items tracked
  Week 1 | 0.84 (0.06) | 0.82 (0.07) | 0.82 (0.06) | 0.84 (0.07)
  Week 2 | 0.71 (0.09) | 0.68 (0.09) | 0.68 (0.09) | 0.71 (0.09)
  Week 3 | 0.69 (0.09) | 0.61 (0.09) | 0.64 (0.09) | 0.66 (0.09)
  Week 4 | 0.67 (0.12) | 0.52 (0.13) | 0.59 (0.12) | 0.59 (0.13)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise vs No Gamification vs Gamification; A standard alpha level of ≥ 0.05 was used to determine statistical significance; Test type: Other; p = 0.01, ANOVA; Linear mixed-factor ANOVA was used with between-subject factors of praise and gamification status, a within-subject factor of time (week), and a dependent variable of DSM timing (Proportion of Items Tracked on Day of Intake). Results reflect outcomes for main effect of time

5. Primary Outcome: Number of Logging Sessions, Overall
Description: The average number of logging sessions per day. Sessions were considered distinct tracking events if they occurred >15 minutes apart.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: logging sessions/day
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
logging sessions/day | 24.6 (2.8) | 21.5 (2.9) | 22.4 (2.8) | 23.7 (2.9)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise; A standard alpha level of ≥ 0.05 was used to determine statistical significance; Test type: Other; p > 0.05, ANOVA; To determine the main effects of positive reinforcement on DSM behavior, a 2x2 factorial ANOVA was conducted with gamification and caregiver praise status as the independent variables and a dependent variable of DSM timing (number of logging sessions). A gamification*caregiver praise interaction term was also included in the model to test for interactive effects
Statistical Analysis 2: Comparison: No Gamification vs Gamification; Test type: Other; p > 0.05, ANOVA; [other analysis details as in outcome 5, analysis 1]

6. Primary Outcome: Number of Logging Sessions, Weekly
Description: as for outcome 5
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: logging sessions/day
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
logging sessions/day
  Week 1 | 7.0 (0.6) | 7.2 (0.7) | 7.1 (0.6) | 7.1 (0.7)
  Week 2 | 8.1 (1.2) | 5.2 (1.3) | 7.2 (1.2) | 6.1 (1.3)
  Week 3 | 5.0 (0.8) | 5.6 (0.9) | 5.0 (0.8) | 5.6 (0.9)
  Week 4 | 4.5 (0.7) | 3.3 (0.7) | 3.1 (0.7) | 4.7 (0.7)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise vs No Gamification vs Gamification; A standard alpha level of ≥ 0.05 was used to determine statistical significance; Test type: Other; p < 0.0001, ANOVA; Linear mixed-factor ANOVA was used with between-subject factors of praise and gamification status, a within-subject factor of time (week), and a dependent variable of DSM timing (number of loging sessions). Results reflect outcomes for main effect of time

7. Secondary Outcome: Child Intrinsic Motivation
Description: Gamification and caregiver praise may differentially affect child motivation to engage in DSM. The Task Evaluation Questionnaire of the Intrinsic Motivation Inventory (IMI) was used to determine whether there were differences in pre-post changes in child intrinsic motivation. This questionnaire consists of 22 items and utilizes a 5-point Likert scale (not at all true to very true) to assess interest/enjoyment, perceived choice, perceived competence, and pressure/tension. At baseline, the measure was administered after the child has practiced using the log with the research assistant so that he or she had some familiarity with the behavior before completing the measure.
  Scales range from 1 to 7, with a higher score indicating a greater degree of the respective motivation subdomain.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
Units on a scale
  Interest/enjoyment | 4.7 (0.6) | 3.9 (0.6) | 3.3 (0.6) | 5.2 (0.6)
  Perceived competence | 5.4 (0.4) | 4.7 (0.5) | 4.4 (0.4) | 5.6 (0.4)
  Perceived choice | 4.8 (0.4) | 5.5 (0.4) | 5.4 (0.4) | 4.8 (0.4)
  Pressure/tension | 1.8 (0.3) | 3.5 (0.3) | 1.9 (0.3) | 2.4 (0.3)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise; Test type: Other; p > 0.05, ANCOVA; To determine the main effects of positive reinforcement on motivation, a 2x2 factorial ANCOVA was conducted with gamification and caregiver praise status as the independent variables, a dependent variable of intrinsic motivation at follow-up, and a covariate of intrinsic motivation at baseline. A gamification*caregiver praise interaction term was also included in the model to test for interactive effects
Statistical Analysis 2: Comparison: No Gamification vs Gamification; Test type: Other; p > 0.05, ANCOVA; [other analysis details as in outcome 7, analysis 1]

8. Secondary Outcome: Child Motivation to Change Eating Behaviors
Description: Child's motivation to change eating habits will be measured, as this may influence engagement in DSM. Children will be asked to complete the 8-item diet subscale of the Motivation to Exercise and Diet Questionnaire-Adapted for Children (MED-C), which is based on self-determination theory. The MED-C diet subscale utilizes a 5-point Likert scale (never to always) and includes 5 items related to motivation and 3 items related to self-determination theory needs (autonomy, competence, relatedness). This validity of the questionnaire has been tested in children aged 7 to 11 years.
  Scale ranges from 0 to 32, with a higher score indicating greater motivation to change eating habits.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
Units on a scale | 30.9 (0.7) | 30.4 (0.8) | 30.1 (0.7) | 31.2 (0.8)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise; A standard alpha level of ≥ 0.05 was used to determine statistical significance; Test type: Other; p > 0.05, ANCOVA; To determine the main effects of positive reinforcement on motivation, a 2x2 factorial ANCOVA was conducted with gamification and caregiver praise status as the independent variables, a dependent variable of scores for child motivation to change eating behaviors at follow-up, and a covariate of baseline scores. A gamification*caregiver praise interaction term was also included in the model to test for interactive effects
Statistical Analysis 2: Comparison: No Gamification vs Gamification; Test type: Other; p > 0.05, ANCOVA; [other analysis details as in outcome 8, analysis 1]

9. Secondary Outcome: Child Dietary Intake, Fruit
Description: The act of self-monitoring a behavior may result in reactivity, or improvements in the monitored behavior in the absence of other intervention. Thus, child dietary intake will also be assessed at baseline and follow-up using the Block Food Screener for Ages 2-17 2007. The instrument asks about intake in the "last week" and focuses on take of fruit, fruit juices, vegetables, potatoes (including French fries), whole grains, animal-based proteins, dairy, legumes, saturated fat, added sugars (in sweetened cereals, sugar sweetened beverages), glycemic load and glycemic index. It takes approximately 10-12 minutes to complete.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cup equivalents
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
cup equivalents | 1.2 (0.2) | 0.9 (0.2) | 0.9 (0.2) | 1.2 (0.2)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise; Test type: Other; p > 0.05, ANCOVA; To determine the main effects of positive reinforcement on dietary intake, a 2x2 factorial ANCOVA was conducted with gamification and caregiver praise status as the independent variables, a dietary intake at follow-up, and a covariate of dietary intake at baseline. A gamification*caregiver praise interaction term was also included in the model to test for interactive effects
Statistical Analysis 2: Comparison: No Gamification vs Gamification; A standard alpha level of ≥ 0.05 was used to determine statistical significance; Test type: Other; p > 0.05, ANCOVA; [other analysis details as in outcome 9, analysis 1]

10. Secondary Outcome: Child Dietary Intake, Vegetables Excluding Potatoes
Description: as for outcome 9
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cup equivalents
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
cup equivalents | .6 (.1) | .6 (.1) | .4 (.1) | .8 (.1)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise; A standard alpha level of ≥ 0.05 was used to determine statistical significance; Test type: Other; p > 0.05, ANCOVA; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: No Gamification vs Gamification; Test type: Other; p = 0.03, ANCOVA; [other analysis details as in outcome 9, analysis 1]

11. Secondary Outcome: Child Dietary Intake, Potatoes
Description: as for outcome 9
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cup equivalents
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
cup equivalents | .2 (.04) | .2 (.04) | .1 (.03) | .3 (.04)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise; Test type: Other; p > 0.05, ANCOVA; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: No Gamification vs Gamification; Test type: Other; p = 0.02, ANCOVA; [other analysis details as in outcome 9, analysis 1]

12. Secondary Outcome: Child Dietary Intake, Sweet & Salty Snack Foods
Description: as for outcome 9
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: g
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
g | 36.5 (7.9) | 46.5 (8.4) | 38.3 (8.0) | 44.7 (8.5)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise; Test type: Other; p > 0.05, ANCOVA; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: No Gamification vs Gamification; Test type: Other; p > 0.05, ANCOVA; [other analysis details as in outcome 9, analysis 1]

13. Secondary Outcome: Child Dietary Intake, Sugar-sweetened Beverages
Description: as for outcome 9
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kilocalories
Arm/Group | No Caregiver Praise | Caregiver Praise | No Gamification | Gamification
Number analyzed (Participants) | 10 | 9 | 10 | 9
kilocalories | 28.1 (7.8) | 26.0 (8.2) | 33.2 (7.7) | 20.9 (8.2)
Statistical Analysis 1: Comparison: No Caregiver Praise vs Caregiver Praise; Test type: Other; p > 0.05, ANCOVA; [other analysis details as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: No Gamification vs Gamification; Test type: Other; p > 0.05, ANCOVA; [other analysis details as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Children: BASIC; Parent: BASIC: Children will be asked to track their intake of fruits, vegetables, sweet and salty snack foods, and sugary drinks in the web-based dietary self-monitoring (DSM) log for 4 weeks. Each child will be provided with a personal URL to access their log, which can be accessed from any internet-capable device (computer, phone, etc.). Caregivers will be asked to review their child's log each day and complete a caregiver check-in in the DSM log.
- Children: PRAISE; Parent: PRAISE: In addition to conditions of the BASIC group, caregivers will also be asked to provide praise to their child for engaging in DSM over the 4 weeks. Additionally, when the caregiver completes caregiver check-ins in the DSM log, they will receive a prompt to also complete a praise check-in.
  Caregiver Praise: Caregivers will provide praise for child's engagement in dietary self-monitoring behaviors as a form of positive reinforcement
- Children: GAME; Parent: GAME: In addition to the conditions of the BASIC group, the child's log will also include a virtual pet that evolves over time as he/she uses the log. As the child earns points, the pet will level up and grow over time.
  Gamification: DSM logs will include gamification (points, levels, virtual pets) as positive reinforcement for child's engagement in dietary self-monitoring behaviors
- Children: PRAISE+GAME; Parent: PRAISE+GAME: In addition to conditions of the BASIC group, caregivers will also be asked to provide praise to their child for engaging in DSM over the 4 weeks. Additionally, when the caregiver completes caregiver check-ins in the DSM log, they will receive a prompt to also complete a praise check-in. The child's log will also include a virtual pet that evolves over time as he/she uses the log. As the child earns points, the pet will level up and grow over time.
  Caregiver Praise: Caregivers will provide praise for child's engagement in dietary self-monitoring behaviors as a form of positive reinforcement
  Gamification: DSM logs will include gamification (points, levels, virtual pets) as positive reinforcement for child's engagement in dietary self-monitoring behaviors
Arm/Group | Children: BASIC | Children: PRAISE | Children: GAME | Children: PRAISE+GAME | Parent: BASIC | Parent: PRAISE | Parent: GAME | Parent: PRAISE+GAME
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/4 | 0/5 | 0/5 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/4 | 0/5 | 0/5 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/4 | 0/5 | 0/5 | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT06193967/Prot_SAP_002.pdf
  • Informed Consent Form (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT06193967/ICF_003.pdf